CLINICAL TRIAL: NCT03362177
Title: RECITE: A Phase 3 Randomized Placebo-controlled Double-blind Study of Romiplostim for the Treatment of Chemotherapy- Induced Thrombocytopenia in Patients Receiving Oxaliplatin-based Chemotherapy for Treatment of Gastrointestinal, Pancreatic, or Colorectal Cancer
Brief Title: Study of Romiplostim for Chemotherapy-induced Thrombocytopenia in Adult Subjects With Gastrointestinal, Pancreatic, or Colorectal Cancer
Acronym: RECITE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20140346; 2017-002992-25 (EudraCT Number)
Record Dates: First submitted 2017-10-12; First posted 2017-12-05 (Actual); Results first posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Chemotherapy-induced Thrombocytopenia
Keywords: Chemotherapy Induced Thrombocytopenia; Gastrointestinal Cancer; Colorectal Cancer; Pancreatic Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms; Colorectal Neoplasms; Pancreatic Neoplasms | interventions — romiplostim

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Romiplostim (Experimental): Participants will be enrolled to the study in a 2:1 randomization ratio. Amgen investigational product (romiplostim or placebo) will be administered in the clinic by a qualified healthcare provider as a subcutaneous injection.
  Interventions: Biological: Romiplostim
- Placebo (Placebo Comparator): Participants will be enrolled to the study in a 2:1 randomization ratio. Amgen investigational product (romiplostim or placebo) will be administered in the clinic by a qualified healthcare provider as a subcutaneous injection.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Romiplostim — This study is designed to study Romiplostim for the treatment of chemotherapy-induced thrombocytopenia (CIT) in patients receiving chemotherapy for the treatment of gastrointestinal/colorectal/pancreatic cancer.
  Arms: Romiplostim
Other: Placebo — Placebo Comparator
  Arms: Placebo

SUMMARY:
Study of Romiplostim for Chemotherapy-induced Thrombocytopenia in Adult Subjects with Gastrointestinal, Pancreatic, or Colorectal Cancer

DETAILED DESCRIPTION:
RECITE: A phase 3 Randomized Placebo-controlled Double-blind Study of Romiplostim for the Treatment of Chemotherapy-induced Thrombocytopenia in Patients Receiving Oxaliplatin-based Chemotherapy for Treatment of Gastrointestinal, Pancreatic, or Colorectal Cancer

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent prior to initiation of any study specific activities/procedures or subject's legally acceptable representative has provided informed consent prior to any study-specific activities/procedures being initiated when the subject has any kind of condition that, in the opinion of the investigator, may compromise the ability of the subject to give written informed consent.
* Males or females greater than or equal to 18 years of age at signing of the informed consent.
* Histologically or cytologically confirmed diagnosis of gastrointestinal, pancreatic, or colorectal adenocarcinoma, defined as cancers of the esophagus (including esophagogastric junction [EGJ] cancer), stomach, pancreas, colon, or rectum. Tumor stage will not affect eligibility.
* Subjects must be receiving 1 of the following regimens: An oxaliplatin-based chemotherapy regimen, containing 5 FU or capecitabine plus oxaliplatin (irinotecan may be added for FOLFIRINOX or FOLFOXIRI) on a 14- or 21 day schedule, respectively; OR, subjects must have chemotherapy-induced thrombocytopenia from a non-protocol chemotherapy regimen, planning to start treatment with one of the protocol chemotherapy regimens which has been delayed greater than or equal to one week due to chemotherapy-induced thrombocytopenia. Note: Use of these regimens are permitted with (1) anti angiogenic agents (such as bevacizumab) or (2) targeted therapy (such as anti epidermal growth factor receptor agents);
* Subjects must have a local platelet count ≤ 85 x 10^9/L on study day 1.
* Subjects must be at least 14 days removed from the start of the chemotherapy cycle immediately prior to study day 1 if they received FOLFOX, FOLFIRINOX or FOLFOXIRI, and 21 days removed if they received CAPEOX.
* Subjects must have at least 3 remaining planned cycles of chemotherapy at study enrollment.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.

Exclusion Criteria:

Previous or Current Medical Conditions

* Acute lymphoblastic leukemia.
* Acute myeloid leukemia.
* Any myeloid malignancy.
* Myelodysplastic syndrome. Baseline bone marrow biopsy is not required to rule out MDS. However, if a bone marrow biopsy and cytogenetics were performed as part of diagnostic or staging work-up, these results will be collected to confirm.
* Myeloproliferative disease.
* Multiple myeloma.
* Within 4 months prior to enrollment, any history of active congestive heart failure (New York Heart Association [NYHA] Class III to IV), symptomatic ischemia, uncontrolled arrhythmias, clinically significant electrocardiogram (ECG) abnormalities, screening ECG with corrected QT (QTc) interval of > 470 msec, pericardial disease, or myocardial infarction.
* Major surgery ≤ 28 days or minor surgery ≤ 3 days prior to enrollment.
* New or uncontrolled venous thromboembolism or thrombotic events within 3 months prior to screening. To be eligible, subjects must have received at least 14 days of anticoagulation for a new thrombotic event and considered to be both stable and suitable for continued therapeutic anticoagulation during trial participation.
* History of arterial thrombosis (eg, stroke or transient ischemic attack) within 6 months of screening.
* Evidence of active infection within 2 weeks prior to first dose of study treatment.
* Known human immunodeficiency virus infection. Subjects without a documented diagnosis in their medical history will require a local laboratory assessment at screening. If local laboratory results are not available, use central laboratory results.
* Known active chronic hepatitis B or C infection. Subjects without a documented diagnosis in their medical history will require a local laboratory assessment at screening. If local laboratory results are not available, use central laboratory results. Hepatitis B and C infection is based on the following results:
* Positive for hepatitis B surface antigen (HBsAg) (indicative of chronic hepatitis B or recent acute hepatitis B).
* Negative HBsAg and positive for hepatitis B core antibody: hepatitis B virus DNA by polymerase chain reaction (PCR) is necessary. Detectable hepatitis B virus DNA suggests occult hepatitis B.
* Positive Hepatitis C virus antibody (HCVAb): hepatitis C virus RNA by PCR is necessary. Detectable hepatitis C virus RNA suggests chronic hepatitis C.
* Secondary malignancy within the past 5 years except:
* Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
* Adequately treated cervical carcinoma in situ without evidence of disease.
* Adequately treated breast ductal carcinoma in situ without evidence of disease.
* Prostatic intraepithelial neoplasia without evidence of prostate cancer.
* Adequately treated urothelial papillary noninvasive carcinoma or carcinoma in situ.
* Malignancy treated with curative intent and with no known active disease present for at least 3 years before enrollment and felt to be at low risk for recurrence by the treating physician
* Thrombocytopenia due to another etiology other than CIT (eg, chronic liver disease, prior history of immune thrombocytopenia purpura).

Prior/Concomitant Therapy

• Previous use of romiplostim, pegylated recombinant human megakaryocyte growth and development factor, eltrombopag, recombinant human TPO, any other TPO receptor agonist, or any investigational platelet producing agent.

Prior/Concurrent Clinical Study Experience • Currently receiving treatment in another investigational device or drug study, or less than 28 days since ending treatment on another investigational device or drug study(ies). Other investigational procedures while participating in this study are excluded.

Diagnostic Assessments

* Anemia (hemoglobin <80 g/L [8 g/dL]) on the day of initiation of investigational product as assessed by local labs. Use of red cell transfusions and erythropoietic stimulating agents is permitted throughout the study as per institutional guidelines.
* Neutropenia (absolute neutrophil count 1 x 10^9/L) on the day of initiation of investigational product as assessed by local labs. Use of granulocyte-colony stimulating factor is permitted throughout the study as per institutional guidelines.
* Abnormal renal function with creatinine clearance < 30 mL/min using the Cockcroft-Gault estimated creatinine clearance as assessed by local laboratory during screening. If local laboratory results are not available, use central laboratory results.
* Abnormal liver function (total bilirubin > 3 X ULN; alanine aminotransferase [ALT] or aspartate aminotransferase [AST] > 3 X ULN for subjects without liver metastases or ≥ 5 X ULN for subjects with liver metastases) as assessed by local laboratory during screening. If local laboratory results are not available, use central laboratory results.

Other Exclusions

* Females who are pregnant or breastfeeding or planning to become pregnant or breastfeed during treatment and for an additional 6 months after treatment (and chemotherapy) discontinuation (females of childbearing potential should only be included after a confirmed menstrual period and a negative highly sensitive urine or serum pregnancy test.)
* Females of childbearing potential unwilling to use a highly effective method of contraception during treatment and for an additional 6 months after treatment (and chemotherapy) discontinuation.
* Males unwilling to use contraception* (male condom or sexual abstinence) or their female partner(s) of childbearing potential who are unwilling to use a highly effective method of contraception during treatment (and chemotherapy) and for an additional 6 months after treatment (and chemotherapy) discontinuation.

  *If the male's sole partner is of non-childbearing potential, he is not required to use additional forms of contraception during the study.
* Subject has known sensitivity to any of the products to be administered during dosing.
* Subject likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures (eg, COAs) to the best of the subject and investigator's knowledge.
* History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.
* Male subjects with a pregnant partner who are unwilling to practice abstinence or use a condom during treatment (and chemotherapy) and for an additional period of 6 months after treatment (and chemotherapy) discontinuation.
* Male subjects unwilling to abstain from donating sperm during treatment (and chemotherapy) and for an additional 6 months after treatment (and chemotherapy) discontinuation.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2025-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (116):
- United States (22):
  - Saint Bernards Medical Center, Jonesboro, Arkansas
  - Pacific Cancer Medical Center Inc, Anaheim, California
  - University of California Irvine, Orange, California
  - Colorado West Healthcare System dba Grand Valley Oncology, Grand Junction, Colorado
  - Mid Florida Hematology and Oncology Centers PA, Orange City, Florida
  - Oncology and Hematology Associates of West Broward, PA, Tamarac, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Orchard Healthcare Research Inc, Skokie, Illinois
  - Christus Saint Frances Cabrini Hospital, Alexandria, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Christus Highland Cancer Treatment Center, Shreveport, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - American Oncology Partners, PA, Bethesda, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Hattiesburg Clinic Hematology/Oncology, Hattiesburg, Mississippi
  - Oncology Hematology Associates, Springfield, Missouri
  - Morristown Medical Center, Morristown, New Jersey
  - Regional Cancer Care Associates, Sparta, New Jersey
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Medical Oncology Associates PS, Spokane, Washington
  - Yakima Valley Memorial Hospital, Yakima, Washington
- Argentina (4):
  - Hospital Universitario Fundacion Favaloro, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Instituto Oncologico Cordoba, Córdoba, Córdoba Province
  - Centro de Investigaciones Clínicas Clínica Viedma, Viedma, Río Negro Province
  - Centro de Diagnostico Investigacion y Tratamiento, Salta
- Austria (2):
  - Landeskrankenhaus Steyr, Steyr
  - Universitaetsklinikum Allgemeines Krankenhaus Wien, Vienna
- Brazil (6):
  - Instituto de Oncologia do Parana, Curitiba, Paraná
  - Vencer e Oncoclinica, Teresina, Piauí
  - Centro de Pesquisa da Serra Gaucha - Cepesg, Caxias do Sul, Rio Grande do Sul
  - Catarina Pesquisa Clinica, Itajaí, Santa Catarina
  - Loema Instituto de Pesquisa Clinica e Consultores Ltda, Campinas, São Paulo
  - Casa de Saude Santa Marcelina, São Paulo, São Paulo
- Bulgaria (3):
  - Complex Oncology Center - Ruse EOOD, Rousse
  - Medical Center Nadezhda Clinical EOOD, Sofia
  - Specialized Hospital for Active Treatment of Oncology EAD, Sofia
- Canada (2):
  - Cape Breton Cancer Centre, Nova Scotia Health Authority, Sydney, Nova Scotia
  - Grand River Regional Cancer Centre at Grand River Hospital, Kitchener, Ontario
- Colombia (3):
  - Fundacion Colombiana de Cancerologia Clinica Vida, Medellín, Antioquia
  - Oncomedica Imat, Montería, Departamento de Córdoba
  - Centro Medico Imbanaco, Cali, Valle del Cauca Department
- France (4):
  - Centre Hospitalier Universitaire de Brest, Brest
  - Hôpital Européen Georges Pompidou, Paris
  - Hopital Foch, Suresnes
  - Institut Gustave Roussy, Villejuif
- Greece (7):
  - General Hospital of Athens Laiko, Athens
  - Aretaieio Hospital, Athens
  - Evgenidio Hospital I Agia Trias, Athens
  - Attikon University Hospital, Athens
  - General Oncology Hospital of Kifissia Agioi Anargyroi, Athens
  - University Hospital of Patras, Pátrai
  - Agios Loukas Clinic, Thessaloniki
- Hungary (4):
  - Del-pesti Centrumkorhaz - Orszagos Hematologiai es Infektologiai Intezet, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Gyor-Moson-Sopron Varmegyei Petz Aladar Egyetemi Oktatokorhaz, Győr
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont Altalanos Orvostudomanyi Kar, Szeged
- Italy (3):
  - Azienda Socio Sanitaria Territoriale di Cremona, Cremona
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliera Citta della Salute e della Scienza di Torino Ospedale Molinette, Torino
- Mexico (4):
  - Oncotech, La Paz, Baja California Sur
  - Centro de Atencion e Investigacion Cardiovascular del Potosi Sc, San Luis Potosí City, San Luis Potosí
  - Centro Medico Nacional Siglo XXI, México
  - Oaxaca Site Management Organization SC, Oaxaca City
- Peru (2):
  - Hospital Goyeneche, Arequipa
  - Oncosalud, Lima
- Poland (3):
  - Wojewodzki Szpital Specjalistyczny w Bialej Podlaskiej, Biała Podlaska
  - Powiatowe Centrum Zdrowia w Brzezinach Sp Z o o, Brzeziny
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Poznan
- Portugal (5):
  - Centro Hospitalar Universitario de Lisboa Norte, EPE - Hospital de Santa Maria, Lisbon
  - Unidade Local de Saude de Matosinhos, EPE - Hospital Pedro Hispano, Matosinhos Municipality
  - Centro Hospitalar Universitario do Porto, EPE - Hospital de Santo Antonio, Porto
  - Centro Hospitalar Universitario de Sao Joao, EPE - Hospital Sao Joao, Porto
  - Centro Hospitalar Tras-os-Montes e Alto Douro EPE - Unidade de Vila Real, Vila Real
- Romania (7):
  - Policlinica de Diagnostic Rapid, Brasov
  - Fundeni Clinical Institute for Digestive Disorders and Liver Transplantation, Bucharest
  - Spitalul Clinic al Cailor Ferate Cluj Napoca, Cluj-Napoca
  - SC Medisprof SRL, Cluj-Napoca
  - Centrul de Oncologie Sf Nectarie SRL, Craiova
  - Institutul Regional de Oncologie Iasi, Iași
  - SC Oncomed SRL, Timișoara
- Russia (13):
  - SBHI of Arkhangelsk region Arkhangelsk clinical oncology dispensary, Arkhangelsk
  - Autonomic SHI Republican clinical oncology dispensary of MoH of the Republic of Tatarstan, Kazan'
  - Clinical hospital 2, Group of companies medsi, Moscow
  - Medsi Group, Moscow Region
  - LLC Tonus, Nizhny Novgorod
  - Omsk Regional Clinical Oncology Dispensary, Omsk
  - State budget institution of public health Pyatigorsk oncology dispensary, Pyatigorsk
  - State Institution of Public Health, Ryazan
  - Leningrad Regional Oncology Dispensary na L D Roman, Saint Petersburg
  - FSBI Scientific and Research Oncology Institute named after N N Petrov, Saint Petersburg
  - State Institution of Public Health Oncology Dispensary 2 of Public Health Krasnodar Region, Sochi
  - State Institution of Public Health Tambov Regional Oncology Dispensary, Tambov
  - Respublican clinical oncology dispensary Minzdrava of Republic of Bashkortostan, Ufa
- Spain (6):
  - Hospital Clinico Universitario San Cecilio, Granada, Andalusia
  - Hospital Clinico Universitario de Salamanca, Salamanca, Castille and León
  - Hospital Universitario Arnau de Vilanova Lleida, Lleida, Catalonia
  - Hospital Universitari Sant Joan de Reus, Reus, Catalonia
  - Complexo Hospitalario Universitario de Ourense, Ourense, Galicia
  - Hospital Universitario Madrid Sanchinarro, Madrid
- Turkey (Türkiye) (13):
  - Baskent Universitesi Adana Doktor Turgut Noyan Uygulama ve Arastirma Merkezi, Adana
  - Doktor Abdurrahman Yurtaslan Ankara Onkoloji Egitim ve Arastirma Hastanesi, Ankara
  - Hacettepe Universitesi Tip Fakultesi, Ankara
  - Gazi Universitesi Saglik Arastirma ve Uygulama Merkezi Gazi Hastanesi, Ankara
  - Ankara Bilkent Sehir Hastanesi, Ankara
  - Trakya Universitesi Saglik Arastirma ve Uygulama Merkezi, Edirne
  - Istanbul Universitesi Onkoloji Enstitusu, Istanbul
  - Prof Dr Cemil Tascioglu Sehir Hastanesi, Istanbul
  - Goztepe Prof Dr Suleyman Yalcin Sehir Hastanesi, Istanbul
  - Ege Universitesi Tip Fakultesi, Izmir
  - Izmir Ekonomi Universitesi Medical Point Hastanesi, Izmir
  - Kocaeli Universitesi Arastirma ve Uygulama Hastanesi, Kocaeli
  - VM Medical Park Samsun Hastanesi, Samsun
- Ukraine (3):
  - Communal Institution Chernivtsi Regional Clinical Oncological Dispensary, Chernivtsi
  - Prykarpatskyy Clinical Oncology Centre, Ivano-Frankivsk
  - Transcarpathian Regional Clinical Oncological Dispensary, Uzhhorod

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in 55 trial centers in Bulgaria, Greece, Italy, Poland, Portugal, Romania, Spain, Argentina, Brazil, Canada, Mexico, Russia, Turkey, and the United States.
Pre-assignment Details: Adult participants receiving oxaliplatin-based chemotherapy regimens for the treatment of gastrointestinal, pancreatic, or colorectal adenocarcinoma were enrolled. Participants were randomized in a 2:1 ratio to receive either romiplostim or placebo, respectively. Randomization was stratified by tumor type and baseline platelet count (<50 x 10^9/L and ≥ 50 x 10^9/L).
Groups:
- Romiplostim: Participants were randomized to receive weekly subcutaneous (SC) injections of romiplostim for up to 21 weeks.
  Doses started at 2mcg/kg of body weight and increased by increments of 1 mcg/kg to a maximum dose of 10 mcg/kg, or until a target platelet count of ≥ 100 x 10^9/L.
  Participants continued to receive oxaliplatin-based chemotherapy in cycles of up to 3 weeks duration.
  Following the last dose of romiplostim, participants remained in the long-term follow-up period for up to 1 year.
- Placebo: Participants were randomized to receive weekly SC injections of placebo for up to 21 weeks.
  Participants' platelet levels were monitored throughout the treatment period. Participants continued to receive oxaliplatin-based chemotherapy in cycles of up to 3 weeks duration.
  Following the last dose of placebo, participants remained in the long-term follow-up period for up to 1 year.
Period: Overall Study
Arm/Group | Romiplostim | Placebo
Started | 109 | 56
Safety Analysis Set (Included all randomized participants who received at least 1 dose of investigational product, according to actual treatment received.) | 110 (One participant randomized to the placebo group received romiplostim.) | 55
Completed | 34 | 26
Not Completed | 75 | 30
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 12 | 8
Not completed — Decision by sponsor | 6 | 0
Not completed — Death | 55 | 22

BASELINE CHARACTERISTICS:
Groups:
- Romiplostim: Participants were randomized to receive weekly SC injections of romiplostim for up to 21 weeks.
  Doses started at 2mcg/kg of body weight and increased by increments of 1 mcg/kg to a maximum dose of 10 mcg/kg, or until a target platelet count of ≥ 100 x 10^9/L.
  Participants continued to receive oxaliplatin-based chemotherapy in cycles of up to 3 weeks duration.
  Following the last dose of romiplostim, participants remained in the long-term follow-up period for up to 1 year.
- Total: Total of all reporting groups
Arm/Group | Romiplostim | Placebo | Total
Number analyzed (Participants) | 109 | 56 | 165
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 57 | 33 | 90
  >=65 years | 52 | 23 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (10.9) | 60.9 (11.5) | 61.4 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 20 | 66
  Male | 63 | 36 | 99
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 11 | 39
  Not Hispanic or Latino | 81 | 45 | 126
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black (or African American) | 4 | 2 | 6
  White | 94 | 54 | 148
  Other | 11 | 0 | 11
Mean Baseline Platelet Count [Mean (Standard Deviation); unit: 10^9 platelets per L] | 67.073 (13.668) | 63.989 (14.709) | 66.027 (14.062)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Had Thrombocytopenia-induced Dose Modification
Description: Participants met the criteria of the primary endpoint if there was no thrombocytopenia-induced modification of any myelosuppressive treatment agent in the second and third cycles of the planned on-trial chemotherapy regimen (cycles were up to 3 weeks).
  A thrombocytopenia-induced modification was defined as any dose reduction, dose delay, dose omission, and/or early chemotherapy treatment discontinuation due to low platelet counts less than 100 x 10^9/L.
  The 95% confidence interval (CI) is based on the exact Clopper-Pearson method.
Time Frame: Day 1 up to Week 12
Population: The full analysis set included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Romiplostim | Placebo
Number analyzed (Participants) | 109 | 56
percentage of participants | 84.4 [76.21 to 90.64] | 35.7 [23.36 to 49.64]
Statistical Analysis 1: Comparison: Romiplostim vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-value was from the stratified exact test of null hypothesis: common treatment odds ratio=1; Odds Ratio (OR) = 10.16, 95% CI 2-sided [4.44 to 23.72] — Odds ratio (romiplostim/placebo) was calculated by using two-sided Cochran-Mantel-Haenszel (CMH) tests considering stratification factors (tumor type and baseline platelet count)

2. Secondary Outcome: Platelet Count Nadir at the End of the Treatment Period
Description: The platelet count nadir from the first on-trial chemotherapy through the end of the treatment period is presented. The least squares (LS) mean platelet count nadirs were estimated using a general linear model which included treatment, stratification factors, and the interaction between treatment and the stratification factors (tumor type and baseline platelet count).
Time Frame: Up to 21 weeks
Population: The full analysis set included all randomized participants.
Measure: Least Squares Mean (95% Confidence Interval); unit: 10^9 platelets per L
Arm/Group | Romiplostim | Placebo
Number analyzed (Participants) | 109 | 56
10^9 platelets per L | 77.3 [66.5 to 88.0] | 51.1 [36.4 to 65.8]
Statistical Analysis 1: Comparison: Romiplostim vs Placebo; Test type: Superiority; p = 0.005, General linear model; General linear model included treatment, stratification factors, and the interaction between treatment and the stratification factors; Mean difference = 26.1, 95% CI 2-sided [7.9 to 44.4] — Romiplostim - placebo

3. Secondary Outcome: Kaplan-Meier Estimate of Time to First Platelet Response
Description: Platelet response was defined as achieving a platelet count of ≥ 100 x 10^9/L in the absence of platelet transfusions during the preceding 7 days.
  Participants who did not achieve a response event during the treatment period were censored at their last platelet count assessment up to end of treatment period or at the randomization date if they did not have any post-baseline platelet assessments.
Time Frame: Up to 21 weeks
Population: The full analysis set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Romiplostim | Placebo
Number analyzed (Participants) | 109 | 56
weeks | 1.1 [NA to NA] — The upper and lower 95% CIs of the median were not estimable as no participants were censored or had any events for the interval from the first quarter to the median month (i.e., no variability). | 2.1 [1.1 to 3.0]
Statistical Analysis 1: Comparison: Romiplostim vs Placebo; Test type: Superiority; p < 0.001, Cox proportional hazards; Cox proportional hazards model was stratified by randomization factors (tumor type and baseline platelet count); Hazard Ratio (HR) = 2.673, 95% CI 2-sided [1.808 to 3.952] — Hazard ratio is romiplostim vs. placebo. A value > 1.0 indicates a higher average event rate and shorter time to response for romiplostim relative to placebo

4. Secondary Outcome: Duration-adjusted Event Rate of Bleeding Events in the Treatment Period
Description: The duration-adjusted adverse event (AE) incidence rate was the number of events per 100 subject-years from the trial day 1 until the date of last dose of investigational product + 30 days, or end of trial, whichever is earlier.
  It was calculated as: duration-adjusted event rate per 100 subject years (n/Subj-yr) x 100.
  The duration-adjusted event rate was assessed for Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 Grade 2 bleeding events. CTCAE grading for AEs ranges from Grade 1 (mild) to Grade 5 (death related to AE). Grade 2 AEs were moderate.
Time Frame: Up to 21 weeks
Population: The full analysis set included all randomized participants.
Measure: Number; unit: bleeding events per 100 subject-years
Arm/Group | Romiplostim | Placebo
Number analyzed (Participants) | 109 | 56
bleeding events per 100 subject-years | 4.0 | 7.6
Statistical Analysis 1: Comparison: Romiplostim vs Placebo; Test type: Superiority; p = 0.63, Andersen-Gill model; Andersen-Gill model was stratified by randomization factors (tumor type and baseline platelet count); Hazard Ratio (HR) = 0.53, 95% CI 2-sided [0.04 to 6.77] — Romiplostim/Placebo

5. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time calculated from trial Day 1 to death. Participants who did not died were censored.
Time Frame: From Day 1 up to 1 year after last dose of investigational product (IP) (max 1869 days)
Population: The full analysis set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Romiplostim | Placebo
Number analyzed (Participants) | 109 | 56
months | 21.0 [15.4 to 45.3] | 46.0 [22.2 to NA] — As more than half of the participants were censored, not enough deaths occurred to estimate CI Upper Limit.

6. Secondary Outcome: Percentage of Participants Who Had Platelet Transfusions During the Treatment Period
Description: Participants who had at least 1 platelet transfusion during the treatment period.
Time Frame: Up to 21 weeks
Population: The full analysis set included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Romiplostim | Placebo
Number analyzed (Participants) | 109 | 56
percentage of participants | 1.8 [0.22 to 6.47] | 0.0 [0.00 to 6.38]

7. Secondary Outcome: Percentage of Participants Who Achieved a Platelet Count ≥ 100 x 10^9/L
Description: The number of participants who achieved a platelet count ≥ 100 x 10^9/L at any time after trial Day 1 to Week 4 (7 days after the planned third dose of IP). If a platelet transfusion occurred during the 7 days preceding a platelet count, then that platelet count was not considered as achieving the endpoint even if it is ≥ 100 x 109/L. Participants who had no platelet counts during this period were considered as not achieving achieved a platelet count ≥ 100 x 109/L. For participants who never received IP, the participants are considered as not achieving a platelet count ≥ 100 x 109/L. Weeks with no platelet count measurements (missing data) were considered as not achieving a platelet count ≥ 100 x 109/L.
Time Frame: Day 1 to Week 4
Population: The full analysis set included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Romiplostim | Placebo
Number analyzed (Participants) | 109 | 56
percentage of participants | 96.3 [90.87 to 98.99] | 66.1 [52.19 to 78.19]
Statistical Analysis 1: Comparison: Romiplostim vs Placebo; Test type: Superiority; Odds Ratio (OR) = 16.19, 95% CI 2-sided [4.38 to 88.85]

8. Secondary Outcome: Number of Participants Who Experienced Treatment-emergent Adverse Events (TEAEs), Serious AEs (SAEs) and Fatal AEs
Description: An AE was defined as any untoward medical occurrence in a clinical trial participant.
  A TEAE was an AE that started on or after the first dose of IP up to 30 days after the end of investigational product or last dose of on-trial chemotherapy (up to 3 cycles), whichever occurs later. Clinically significant changes in laboratory values were considered AEs.
  A SAE was defined as any untoward medical occurrence that, met at least 1 ofthe following criteria: resulted in death (fatal), immediately life-threatening,required in-patient hospitalization or prolongation of existing hospitalization,resulted in persistent or significant disability/incapacity or was a congenitalanomaly/birth defect.
Time Frame: From first dose of IP to 30 days after last dose of IP: median (min, max) duration was 86.0 (31.0, 184.0) days
Population: The safety population included all randomized participants who received at least 1 dose of IP. Data is reported according to treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Romiplostim | Placebo
Number analyzed (Participants) | 110 | 55
Participants
  TEAEs | 96 | 34
  SAEs | 23 | 3
  Fatal AEs | 2 | 0

9. Secondary Outcome: Number of Participants Who Developed Anti-romiplostim Antibodies and Anti-thrombopoietin (TPO) Antibodies
Description: Blood samples were collected from all participants for the measurement of anti-romiplostim and anti-TPO binding antibodies. Participants were tested for the presence of anti-romiplostim and anti-TPO antibodies at baseline (pre-existing antibody) and post-baseline (developed antibody). Samples testing positive for binding antibodies were also be tested for neutralizing antibodies.
Time Frame: Up to 21 weeks
Population: The safety population included all randomized participants who received atleast 1 dose of IP. Data is reported according to treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Romiplostim | Placebo
Number analyzed (Participants) | 110 | 55
Participants
  Romiplostim: Binding antibodypositive at or before baseline | 2 | 0
  Romiplostim: Neutralizingantibody positive at or beforebaseline | 0 | 0
  Romiplostim: Binding antibodypositive post-baseline with anegative or no result at baseline | 1 | 0
  Romiplostim: Neutralizingantibody positive post-baselinewith a negative or no result atbaseline | 0 | 0
  TPO: Binding antibody positiveat or before baseline | 0 | 0
  TPO: Neutralizing antibodypositive at or before baseline | 0 | 0
  TPO: Binding antibody positivepost-baseline with a negative orno result at baseline | 1 | 0
  TPO: Neutralizing antibodypositive post-baseline with anegative or no result at baseline | 0 | 0

10. Secondary Outcome: Number of Participants Who Reported Myelodysplastic Syndromes (MDS) and SecondaryMalignancies
Description: Events were identified using narrow search of pre-defined list of preferred terms for myelodysplastic syndromes (SMQ). Secondary malignancies included progression from myelodysplastic syndrome to acute myeloid leukemia (AML).
Time Frame: From Day 1 up to 1 year after last dose of IP (max 1869 days)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Romiplostim | Placebo
Number analyzed (Participants) | 110 | 55
Participants
  MDS | 1 | 0
  Secondary Malignancy | 2 | 3

ADVERSE EVENTS:
Time Frame: For Mortality - From Enrollment to End of trial: median (min, max) time on trial was 529.0 (8.0, 1869.0) days. For TEAEs - From first dose of IP to 30 days after last dose of IP: median (min, max) duration was 86.0 (31.0, 184.0) days.
Description: All-cause mortality is reported for all participants enrolled/randomized in the trial. SAEs and other AEs are reported for all participants who received at least one dose of trial drug. Data is reported according to treatment received.
Groups:
- Placebo; Romiplostim: Participants were randomized to receive weekly SC injections of romiplostim for up to 21 weeks.
  Doses started at 2mcg/kg of body weight and increased by increments of 1 mcg/kg to a maximum dose of 10 mcg/kg, or until a target platelet count of ≥ 100 x 10^9/L.
  Participants continued to receive oxaliplatin-based chemotherapy in cycles of up to 3 weeks duration.
  Following the last dose of romiplostim, participants remained in the long-term follow-up period for up to 1 year.
Arm/Group | Placebo | Romiplostim
All-Cause Mortality (participants affected / at risk) | 25/55 | 58/110
Serious Adverse Events (participants affected / at risk) | 3/55 | 23/110
Other Adverse Events (participants affected / at risk) | 28/55 | 76/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=55) | Romiplostim (N=110)
Anaemia (Blood and lymphatic system disorders) | 0 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 2
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 3
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 2
Respiratory tract infection (Infections and infestations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=55) | Romiplostim (N=110)
Anaemia (Blood and lymphatic system disorders) | 5 | 13
Leukopenia (Blood and lymphatic system disorders) | 1 | 10
Lymphopenia (Blood and lymphatic system disorders) | 1 | 6
Neutropenia (Blood and lymphatic system disorders) | 8 | 21
Thrombocytopenia (Blood and lymphatic system disorders) | 11 | 21
Abdominal pain (Gastrointestinal disorders) | 5 | 8
Diarrhoea (Gastrointestinal disorders) | 4 | 13
Nausea (Gastrointestinal disorders) | 7 | 14
Vomiting (Gastrointestinal disorders) | 4 | 11
Asthenia (General disorders) | 5 | 10
Fatigue (General disorders) | 3 | 11
Decreased appetite (Metabolism and nutrition disorders) | 2 | 7
Neuropathy peripheral (Nervous system disorders) | 5 | 12
Hypertension (Vascular disorders) | 0 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/77/NCT03362177/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-03): https://cdn.clinicaltrials.gov/large-docs/77/NCT03362177/SAP_001.pdf